CLINICAL TRIAL: NCT06792942
Title: Investigation of the Effect of Using "Curtain" as a Distraction Method on Fear, Anxiety and Pain in Diagnostic Procedures Performed in Patients With Suspected Thyroid Mass
Brief Title: Investigation of the Effect of Using "Curtain"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Hamdiye ARDA SÜRÜCÜ, Professor, Dicle University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DICLE-ARDASURUCU-004
Record Dates: First submitted 2025-01-18; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Ultrasound Therapy; Complications; Fine Needle Aspiration Biopsy; Thyroid Nodule (Diagnosis)
Keywords: The curtain; Ultrasound Therapy; Complications; Ultrasound; Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule; Disease

STUDY DESIGN:
Intervention Model Description: fine needle biopsy group and control group
Who Masked: Participant
Masking Description: They do not know the experimental or control procedures that take place
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nature view curtain group (Experimental): During the fine needle biopsy, the patient will look at the nature view curtain on the ceiling.
  Interventions: Other: nature view curtain group
- Control group (No Intervention): patients without of the nature view curtain

INTERVENTIONS:
Other: nature view curtain group — During the fine needle biopsy, the patient will look at the nature view curtain on the ceiling.
  Arms: nature view curtain group

SUMMARY:
Thyroid nodules are among the common health problems in adulthood. Thyroid cancers account for approximately 1% of all malignancies in a year.The majority of cancers are diagnosed by thyroid fine needle aspiration biopsy. The most commonly diagnosed cancer type is papillary thyroid cancer and accounts for 85% of all thyroid cancers.Thyroid Ultrasonography is the most important imaging method used in the evaluation of the thyroid gland and its nodules. It enables the detection of nodules and their characteristics and plays a role in deciding which nodules should be evaluated with fine needle aspiration biopsy.Non-pharmacological treatment methods are interventions that can be used to reduce the side effects of medical, surgical or pharmacological treatments. By using medical treatment and complementary therapy together, nurses can reduce patients' anxiety, support their sleep, create a healing environment and increase their health level.

As a non-pharmacological strategy, distraction can be seen as a cost-effective approach to reduce anxiety in procedures that would cause negative anxiety and increase the opportunity for ease of operation. The curtain method also typically involves the use of visually interesting curtains or partitions that can be drawn around the patient's examination area. These curtains may have calming images or vibrant patterns that can help shift the patient's focus away from the frightening procedure being performed.

DETAILED DESCRIPTION:
Research Type:

It was designed as a randomized controlled experimental study.

Research Population and Sample:

The research sample will consist of patients with suspected thyroid mass who applied to a City Training and Research Hospital. The sample of the study is expected to consist of 100 volunteer patients with suspected thyroid mass who applied to the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of a mass in the thyroid
* No vision problems

Exclusion Criteria:

* Mental health problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Before and after immediately after ultrasound guided fine needle aspiration biopsy procedure
  The scale is used to assess subjectively perceived pain. It is a 10 cm (100 mm) ruler with no pain on one end and the "most severe pain" on the other. The individuals participating in the study are asked to mark the intensity of pain they are currently feeling, explaining that the number "0" on the scale means "I feel no pain" and that the intensity of pain increases as the numbers increase, and the number "10" means" I feel the most severe pain". An increase in the score obtained from the scale in the assessment indicates that the pain is increasing. Each patient will be administered two times.

SECONDARY OUTCOMES:
Fear of Pain Scale-III | Before and after immediately after ultrasound guided fine needle aspiration biopsy procedure
  Fear of Pain Scale-III is a 30-item, 5-point Likert type scale developed to measure fear and/or anxiety about pain. The scale consists of 3 sub-dimensions and there are 10 items in each dimension. Scale items for fear of severe pain are 1, 3, 5, 6, 9,10, 13, 18, 25, 27; scale items for fear of mild pain 2, 4, 7, 12, 19, 22, 23, 24, 28, 30;The scale items for fear of medical pain are 8, 11, 14, 15, 16, 17, 20, 21, 26, 29. In evaluating the score of the scale, which has no inverse expression, the items are rated with a Likert-type scoring ranging from 1 to 5 (1- never, 2-a little, 3-quite a bit,4-a lot, 5-extremely). 1-refers to never feeling fear, 5-expresses excessive fear. The lowest possible score in total is 30 and the highest score is 150. The lowest score that can be obtained for the sub-dimensions is 10 and the highest score is 50. A high score on the scale indicates that the individual's fear of pain is also high.
Beck Anxiety Scale | Before and after immediately after ultrasound guided fine needle aspiration biopsy procedure
  It measures the severity of anxiety symptoms experienced by individuals. Consisting of 21 items, scored between 0-3; It is a scale filled by the patient himself. Score Range is 0-63. Anxiety levels of the patients according to the scores obtained; 0-7 points are classified as no anxiety, 8-15 points as mild anxiety, 16-25 points as moderate anxiety, and 26 and above points as severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Dicle Univertsity, Diyarbakır, South East, Turkey (Türkiye)